CLINICAL TRIAL: NCT00915915
Title: Multicenter, Open-label, Randomized Study to Evaluate Inhibition of Ovulation of Two Transdermal Patch Formulations Containing 0.55 mg Ethinylestradiol and Either 1.05 or 2.1 mg Gestodene in Healthy Young Female Volunteers Over a Period of 3 Treatment Cycles
Brief Title: Inhibition of Ovulation and Pharmacokinetics of Transdermal Ethinylestradiol (EE) and Gestodene (GSD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14348; 2009-009177-10 (EudraCT Number)
Record Dates: First submitted 2009-05-18; First posted 2009-06-08 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Contraception; Ovulation Inhibition
Keywords: Female contraception; Ovulation inhibition
MeSH Terms: interventions — Ethinyl Estradiol; Gestodene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Ethinylestradiol/Gestodene (BAY86-5016)
- Arm 2 (Experimental)
  Interventions: Drug: Ethinylestradiol/Gestodene (BAY86-5016)

INTERVENTIONS:
Drug: Ethinylestradiol/Gestodene (BAY86-5016) — Transdermal patch: 0.55mg Ethinylestradiol (EE+2.1mg GSD)Gestodene; 3x7 days patch- wearing phase and a patch-free interval of 7 days (1 pre-treatment cycle, 3 treatment cycles), 1 Follow - up cycle)
  Arms: Arm 1
Drug: Ethinylestradiol/Gestodene (BAY86-5016) — Transdermal patch: 0.55mg Ethinylestradiol (EE+1.05mg GSD)Gestodene; 3x7 days patch- wearing phase and a patch-free interval of 7 days (1 pre-treatment cycle, 3 treatment cycles), 1 Follow - up cycle)
  Arms: Arm 2

SUMMARY:
Investigation of two transdermal hormone patch formulations for contraception regarding inhibition of ovulation over a period of 3 treatment cycles in healthy young female volunteers

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18 BMI 30 kg/m²
* Healthy female volunteers
* Age 18-35 years (smoker not older than 30 years, inclusive)
* Ovulatory pre-treatment cycle, at least 3 month since delivery
* Abortion or lactation before the first screening examination
* Willingness to use non-hormonal methods of contraception during entire study

Exclusion Criteria:

* Contraindications for use of combined (estrogen/gestodene) contraceptive (e.g. history of venous/artial thromboembolic disease
* Regular intake of medication other than OCs
* Clinically relevant findings (blood pressure, physical and gynaecological examination, laboratory examination) anovulatory pre-treatment cycle

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the proportion of volunteers with ovulation in at least one of the treatment cycles 2 and 3 | 4 months

SECONDARY OUTCOMES:
The primary efficacy variable will be the proportion of volunteers with ovulation in at least one of the treatment cycles 2 and 3 | 4 months
Course of gonadotropins (FSH, LH, P, E2) | 4 months
Endometrial thickness and Follicle size | 4 months
Pharmacokinetics of Ethinylestradiol (EE), Gestodene (GSD) and SHBG in treatment cycles 2 and 3 | 4 Months
Cervical effects (Insler Score) for determination of hormonal effects on the cervix and the cervical mucus during pre-treatment cycle and treatment cycle 3 | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/